CLINICAL TRIAL: NCT07110870
Title: Binaural Beats and Cognitive Physical Dual-task Training for Enhancing Cognitive Function in Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/46
Record Dates: First submitted 2025-04-29; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Elderly; Mild Cognitive Impairment
Keywords: Mid Cognitive Impairment; Elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Binaural Beats with Cognitive Physical Dual task training group (Experimental): It includes participants receiving Binural beats with cognitive-physical dual task training for 08 weeks treatment.
  Interventions: Procedure: Binaural Beats and Cognitive physical dual task training
- Cognitive Physical dual task training group (Experimental): This group involves participants receiving cognitive physical dual task training for a period of 08 weeks.
  Interventions: Procedure: Cognitive Physical Dual task training

INTERVENTIONS:
Procedure: Cognitive Physical Dual task training — Randomized Control Group (A)/ Cognitive Physical Dual Task Training Participants in control group will perform cognitive physical dual task training to improve working memory, attention and executive function in elderly with mild cognitive impairment. Dual-task training involved eight programs consist from simple dual-task to more complex dual-task tasks.
  Cognitive task involves verbal fluency, attention, Forward digit span task, backward digit span task, calculation tasks and memory, aerobic exercise including performing actions like dragging the foot and placing it on floor markers (Marked from 1 to 5), Drawing any letters with their feet while seated, range of motion exercise while standing, forward walking, backward walking, tandem walking and stair climbing and strengthening exercise consisting of Thera-band with low intensity training by arms and by legs and passing/throwing a ball (0.1kg, 0.4kg) will be used for physical tasks. Eight programs will be repeated thrice, resultin
  Arms: Cognitive Physical dual task training group
Procedure: Binaural Beats and Cognitive physical dual task training — In experimental group, Binaural beats will be given 03 min before performing a dual task.
  Participants will be in a quiet room and two tones of different frequencies will be generated through the Audacity Program (Version 3.4.2) via stereo headphones presenting a different tone to each ear.
  Phase-I: A warm-up at the beginning of each session (05 min) with supervised walking exercises on a flat surface.
  Phase II: Binaural beats will be induced thrice a week, for 08 weeks. Alpha, and gamma waves, over 30 min, split into two sub-sessions lasting 12 min each. Participants will be allowed to take a 6-minute rest between sub-sessions. Alpha BB (10 Hz), (R: 410 Hz, L: 400 Hz) and gamma BB (30 Hz) (R: 430 Hz, L: 400 Hz) will be provided.
  Phase-III: Return to calm (05 min) with relaxation and breathing exercises, lying on the floor.
  The stimulus volume, played through stereo headphones will be set by the participants at the start of the session to a comfortably loud level.
  Arms: Binaural Beats with Cognitive Physical Dual task training group

SUMMARY:
Mild cognitive impairment is a typical trasnitional stage betweeen the normal aging process and the onset of dementia. Mental exercises and aerobic exercises can shield brain from cognitive decline in elderly. Cognitive physical dual task training is defined as participation in an activity that requires the person to engage physically and cognitively at the same time. Another approach that can improve cognitive functiom in older adults is binaural beats that can be defined as when two different tones are played into two ears, leading to the perception of a beat at frequency equal to the difference between the two tones.Elderly participants with MCI who meet the inclusion criteria will be selected. The Subjects will be randomly allocated into two groups. One group will receive BB in combination with physical dual-task training while the other group will receive cognitive physical dual-task training only for 8 weeks.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To compare the effects of binaural beats in addition to cognitive-physical dual-task training on working memory in older adults with mild cognitive impairment.
2. To compare the effects of binaural beats in addition to congitive-physical dual-task training on attention in older adults.
3. To compare the effects of binaural beats in addition to cognitive-physical dual-task training executive function in older adults.

HYPOTHESIS:

Alternate Hypothesis:

1. There is statistically significant difference between the group recieving binaural beats combined with cognitive-physical dual-task on working memory capacity compared to the group recieving cognitive-physical dual-task in older adults with MCI.
2. There is statistically significant difference between the group recieving binural beats combined with cognitive-physical dual-task on attention compared to the group recieving cognitive-physical dual-task in older adults with MCI.
3. There is statistically significant difference between the group recieving binural beats combined with cognitive-physical dual-task on executive function compared to the group recieving cognitive-physical dual-task in older adults with MCI.

Null Hypothesis:

1. There is no statistically significant difference between the group recieving binaural beats combined with cognitive-physical dual-task on working memory capacity compared to the group recieving cognitive physical dual-task in older adults with MCI.
2. There is no statistically significant difference between the group recieving binural beats combined with cognitive physical dual-task on attention compared to the group recieving cognitive-physical dual-task in older adults with MCI.
3. There is no statistically significant difference between the group recieving binural beats combined with cognitive physical dual-task on executive function compared to the group recieving cognitive-physical dual-task in older adults with MCI.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Multidisciplinary Lab in FUCP. Study duration: 1 year

Selection Criteria:

Inclusion Criteria

1. Age 55 years and above
2. Male and female both
3. Ability to understand simple instructions.
4. Montreal Cognitive Assessment score from 19-25.

Exclusion Criteria

1. Diagnosed neurological, musculoskeletal, and psychiatric disorders.
2. Participants with diagnosed hearing or vision problems.
3. Participants who take 12 seconds to compelete TUG test.

Technique: Non probability Purposive Sampling

Outcome Measures:

Data will be collected on Demographics and general information. Data will be collected using MOCA, Trail making Test A and B and Digit span test.

Experimental Group (A) = This group will receive Cognitive Physical dual-task training . Their outcomes will be measured at baseline, on 4th,and at 8th week of treatment.

Expermental Group (B) =This group will recive Binural Beats with Cognitive Physical dual-task training outcomes will be measured at baseline, on 4th, and at 8th week of treatment.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study within the community.

A printed questionnaire will be provided to the patients after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

1. While existing literature lacks conclusive evidence of the effectivenss of binaural beats in combination with cognitive- physical dual-task training in older adults with mild cognitive impairment,it is only focused on a single cognitive function rather than a wide range.
2. Furthure past studies have primarily focussed on healthy young adults without any specific condition and potential benefits of binaural beats for this specific population remain largely unexplored.
3. Our study addresses this critical gap in the literature and will provide scientific evidence supporting the efficacy of binural beats in combination with cognitive-physcial dual-task training in older adults with mild cognitive impairmment and their effects on a wider range of cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 55 and above older adults.
* Both male and female.
* Ability to understand simple instructions.
* Montreal Cognitive Assessment score from 19-25.

Exclusion Criteria:

* Diagnosed neurological, musculoskeletal, and psychiatric disorders.
* Participants with diagnosed hearing or vision problems.
* Participants who take ≥12 seconds to complete the TUG test

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Working Memory | 8 weeks
  The Digit Span test is one of the most commonly used measures of immediate working memory. The testing procedure for the Digit Span task will be done according to the standard administration, that is, strings of digits are read to subjects at a rate of 1 per second and the subject is asked to repeat them orally in the correct sequence (either forward or backward). The test is discontinued if the subject fails two consecutive trials. The total score corresponds to the maximum number of digits the subject can repeat correctly.
Attention | 8 weeks
  Montreal cognitive assessment will be used. MoCA is a brief 30-question test that takes around 10-12 minutes to complete. A normal score is regarded to be 26 or higher. A score of 18 to 25 is an indicator of mild cognitive impairment (MCI).
Executive function | 8 weeks
  Trail Making Test (TMT) A and B is a test that measures executive function. TMT is broken into two parts: TMT-A (WM) and TMT-B (EF). Each of the two parts consists of 25 circles scattered across a sheet of paper. Part A contains circles numbered from 1-25, and the individual should connect the numbers by drawing lines in ascending order. Part B contains circles with both numbers (1-13) and letters (A-L); the individual must draw lines to connect the circles in ascending order, with the added challenge of alternating between the numbers and letters (for example, 1-A-2-B-3-C, etc.). Individuals must be encouraged to connect the circles as rapid

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan